CLINICAL TRIAL: NCT02208765
Title: Prognostic Value of Myocardial Perfusion Heterogeneity Assessed by Stress Single Photon Emission Computed Tomography
Brief Title: Prognostic Value of SPECT-imaging Myocardial Perfusion Heterogeneity
Acronym: EVAPERF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 38RC13.723
Record Dates: First submitted 2014-08-04; First posted 2014-08-05 (Estimated); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Coronary Artery Disease; Coronary Atherosclerosis
Keywords: Coronary Circulation; Coronary Artery Disease; Myocardial perfusion imaging; Prognosis
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Study cohort (Other): Any patient referred to the Nuclear Cardiology Laboratory of the University Hospital of Grenoble for myocardial perfusion imaging for diagnosis or prognosis evaluation of suspected or know coronary artery disease
  Interventions: Device: Stress Single Photon Emission Computed Tomography

INTERVENTIONS:
Device: Stress Single Photon Emission Computed Tomography

SUMMARY:
Endothelial dysfunction has been demonstrated to be an early marker of coronary artery disease (CAD). On the other hand, myocardial perfusion single photon emission computed tomography (MP-SPECT) is a widely used technique for evaluation of patients with suspected or known CAD.

Preliminary data suggest that myocardial perfusion heterogeneity (a potential surrogate marker of endothelial dysfunction) can be assessed on conventional MP-SPECT, but its additive and independent prognostic value over the presence of myocardial ischemia remain unknown.

More over, factual data demonstrate that inhalation of particulate matters and gaz (NO2, CO) from air pollution contributes to the development of cardiovascular diseases in the short and long term. The role of air pollution in endothelial dysfunction has been suggested.

Accordingly, the purpose of this study is to evaluate the prognostic value of myocardial perfusion heterogeneity assessed by a new automatized image processing method applied to routine MP-SPECT.

The second purpose is to evaluate the role of air pollution exposure in pathogenesis of cardiovascular disease.

The main hypothesis is that the presence of myocardial perfusion heterogeneity is predictive of 2-year cardiovascular events in patients referred to the Nuclear Cardiology Department for routine evaluation of known or suspected CAD.

The second hypothesis is that microcirculatory coronary dysfunction is a causal link between air pollution and cardiovascular disease.

DETAILED DESCRIPTION:
1. SPECT imaging protocol and analysis Stress tests and SPECTs are performed according to the routine protocols in use in our center. Briefly, at peak stress, patients were injected with thallium-201. Five to 10 minutes after stress, a 5-minutes supine acquisition was performed followed by a 5-minutes prone acquisition. Subsequently, technetium-99m-sestamibi was injected, and 2 minutes later a single 5-minutes rest acquisition was performed. During stress acquisition, patients were imaged in supine and prone positions with their arms positioned over their head. The rest acquisition was only acquired in supine position. The gated SPECT studies were performed at each acquisition. Injected activity (IA) was adjusted for patient weight. For weights of <80 kg/ 80-100 kg/>100 kg, thallium-201 IAs were 74/92/111 MBq and technetium-99m-sestamibi IAs were 300/370/450 MBq, respectively. A uniform imaging pre-treatment for the reconstruction of raw myocardial perfusion imaging data was applied, and images were reconstructed and reoriented to obtain transaxial sections of the left ventricle according to the three standard cardiac planes.
2. In this study, we use a new mathematic technique from entropy analysis to provide precise, objective, automated quantification of perfusion heterogeneity at stress with camera SPECT. This method may be a non-invasive imaging to assess coronary microvascular dysfunction.
3. Air pollution exposure (particule matters and gaz) is estimated by SIRANE dispersion models validated by Air Rhône-Alpes, our regional agency tasked with protecting and managing the ambient air quality. The dispersion models are used to estimate the downwind ambient concentration of air pollutants or toxins emitted from sources such as industrial plants, vehicular traffic or accidental chemical releases.

Air pollution is estimated for each patient thanks to their postal private and professional adresses for different windows of exposure :

* short term windows (2hours to 7 days before the MP-SPECT and cardiovascular events).
* long term windows (1 - 5 years before the MP-SPECT and before cardiovascular events)

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Clinical indication for myocardial perfusion imaging

Exclusion Criteria:

* Pregnancy
* Breast feeding women
* Severe comorbidity with life expectancy 6 months
* Left bundle branch block on ECG making heteogeneity analysis impossible
* Patient not resident in the Rhône-Alpes region

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiac and Cerebrovascular Events (MACCEs) | 2 years
  Composite outcome : cardiac death and/or acute coronary syndrome and/or coronary artery bypass graft and/or percutaneous coronary intervention and/or stroke and/or symptomatic peripheral artery disease

SECONDARY OUTCOMES:
composite secondary outcome : number of cardiac death or nonfatal Myocardial Infarction | 2 years
composite secondary outcome : number of cardiac death or nonfatal Myocardial Infarction or stroke | 2 years
composite secondary outcome : number of participants with myocardial revascularization | 2 years
composite secondary outcome : number of all death or non fatal Myocardial Infarction | 2 years
composite secondary outcome : number of all death or non fatal Myocardial Infarction or non fatal stroke | 2 years
composite secondary outcome : number of all death or non fatal Myocardial Infarction or non fatal stroke or number of participants with myocardial revascularization | 2 years
composite secondary outcome : number of all death or non fatal Myocardial Infarction or non fatal stroke or number of participants with myocardial revascularization or symptomatic peripheral artery disease | 2 years
  peripheral artery disease (intermittent claudication/new episode of critical limb ischaemia, new percutaneous/surgical revascularization, or amputation).
cardiac death | 2 years
  Death from coronary artery disease, heart failure, or sudden death
Non fatal Myocardial Infarction | 2 years
acute coronary syndrome | 2 years
Non fatal Stroke | 2 years
Coronary artery bypass graft and/or percutaneous coronary intervention | 2 years
14 Symptomatic peripheral artery disease (intermittent claudication/new episode of critical limb ischaemia, new percutaneous/surgical revascularization, or amputation) | 2 years
influence of air pollution exposure for short and long terms of exposure on myocardial Heterogeneity Index | inclusion
  Air pollution is estimated for each patient thanks to their postal private and professional adresses for different windows of exposure :
  * short term windows (2hours to 7 days before the MP-SPECT and cardiovascular events).
  * long term windows (1 - 5 years before the MP-SPECT and before cardiovascular events)
influence of air pollution exposure for short and long terms of exposure on cardiovascular events | 2 years
  Air pollution is estimated for each patient thanks to their postal private and professional adresses for different windows of exposure :
  * short term windows (2hours to 7 days before the MP-SPECT and cardiovascular events).
  * long term windows (1 - 5 years before the MP-SPECT and before cardiovascular events)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Vanzetto, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- University Hospital, Grenoble, France

REFERENCES:
- [Background] Verma S, Buchanan MR, Anderson TJ. Endothelial function testing as a biomarker of vascular disease. Circulation. 2003 Oct 28;108(17):2054-9. doi: 10.1161/01.CIR.0000089191.72957.ED. No abstract available. PMID 14581384
- [Background] Schindler TH, Nitzsche EU, Schelbert HR, Olschewski M, Sayre J, Mix M, Brink I, Zhang XL, Kreissl M, Magosaki N, Just H, Solzbach U. Positron emission tomography-measured abnormal responses of myocardial blood flow to sympathetic stimulation are associated with the risk of developing cardiovascular events. J Am Coll Cardiol. 2005 May 3;45(9):1505-12. doi: 10.1016/j.jacc.2005.01.040. PMID 15862426
- [Background] Vanzetto G, Ormezzano O, Fagret D, Comet M, Denis B, Machecourt J. Long-term additive prognostic value of thallium-201 myocardial perfusion imaging over clinical and exercise stress test in low to intermediate risk patients : study in 1137 patients with 6-year follow-up. Circulation. 1999 Oct 5;100(14):1521-7. doi: 10.1161/01.cir.100.14.1521. PMID 10510055
- [Background] Johnson NP, Gould KL. Clinical evaluation of a new concept: resting myocardial perfusion heterogeneity quantified by markovian analysis of PET identifies coronary microvascular dysfunction and early atherosclerosis in 1,034 subjects. J Nucl Med. 2005 Sep;46(9):1427-37. PMID 16157524